CLINICAL TRIAL: NCT04650308
Title: Sex Differences in Neuropeptide Y Serum, But Not in Fat Intake and Body Mass Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Sumatera Utara (Other)
Responsible Party: Principal Investigator, DINA KEUMALA SARI, Principal Investigator, Universitas Sumatera Utara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: USumateraUtara 2
Record Dates: First submitted 2020-11-23; First posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Nutrient Deficiency
Keywords: obesity; appetite; neuropeptide; orexigenic; energy; gender
MeSH Terms: conditions — Obesity; Coitus

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy group (Active Comparator): healthy men and women aged 20-60 years old.
  Interventions: Diagnostic Test: Neuropeptide Y examination
- Non-healthy group (Active Comparator): pregnant women, nursing mothers, impaired kidney and liver function, chronic disease, or other metabolic disorders.
  Interventions: Diagnostic Test: Neuropeptide Y examination

INTERVENTIONS:
Diagnostic Test: Neuropeptide Y examination — This examination was conducted by drawing blood serum from research subjects and performing centrifugation with 2000-3000 revolutions per minute (RPM) for 20 minutes. Furthermore, we carried out blood serum tests to check neuropeptide Y levels using the Human Neuropeptide Y Enzyme-link Immunosorbent Assay (ELISA) kit

SUMMARY:
One's appetite has a role in controlling food intake and maintaining energy balance, but its effect on body metabolism related to obesity is still questionable. The purpose of this study was to determine the levels of neuropeptide Y in healthy people and to see differences in gender and anthropometric parameters. The hypothesis of this study was that there would be differences in neuropeptide Y levels in groups with gender and anthropometric parameter differences.

DETAILED DESCRIPTION:
One's appetite has a role in controlling food intake and maintaining energy balance, but its effect on body metabolism related to obesity is still questionable. The purpose of this study was to determine the levels of neuropeptide Y in healthy people and to see differences in gender and anthropometric parameters. The hypothesis of this study was that there would be differences in neuropeptide Y levels in groups with gender and anthropometric parameter differences. This study was a cross-sectional study involving 62 study subjects, male and female, who did not have chronic diseases or metabolic disorders. This research was conducted from April to September 2020. The parameters examined in this study were neuropeptide Y levels and anthropometric parameters. The statistical analysis performed was the Mann-Whitney test to see the differences between groups. The mean age of the research subjects was 40.48 ± 10.85 years, with the same ethnic distribution. The distribution of men and women was more women than men. Based on anthropometric examination, it was found that obesity nutritional status was more common in the female group than in the male group; however, serum neuropeptide Y levels were found to be significantly different between male and female groups (male group was higher).

ELIGIBILITY:
Inclusion Criteria:

* healthy groups for Neuropeptide Y Serum diagnosis

Exclusion Criteria:

* Non-healthy groups for Neuropeptide Y Serum diagnosis

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 62 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2020-06-17 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
levels of neuropeptide Y | up to 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Universitas Sumatera Utara, Medan, North Sumatra, Indonesia

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-11-18): https://cdn.clinicaltrials.gov/large-docs/08/NCT04650308/Prot_SAP_ICF_000.pdf